CLINICAL TRIAL: NCT01600313
Title: Effect of Low Calorie Diet With Rice Bran Oil on Cardiovascular Risk Factors in Hyperlipidemic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Mostafa Noroozi, Principal investigator, Qazvin University Of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: QUMS-2225
Record Dates: First submitted 2012-05-10; First posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Hyperlipidemias
Keywords: rice bran oil; diet; cardiovascular disease; low density lipoprotein; total cholesterol
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases | interventions — Rice Bran Oil; Tacrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment, control (Experimental)
  Interventions: Dietary Supplement: rice bran oil

INTERVENTIONS:
Dietary Supplement: rice bran oil — Treatment group received the low - calorie diet with(30g/day) rice bran oil
  Other Names: King rice bran oil, Bangkok, Thailand)

SUMMARY:
The purpose of this study is to determine the effect of rice bran oil with low calorie diet on lipid profiles.

DETAILED DESCRIPTION:
This study is parallel groups' randomized clinical trial with a pre and post test design.

The study conducted on hyperglycemia patients who were healthy in other respects and were recruited from nutrition and diet therapy clinic. All subjects received a low calorie diet for 4 weeks from registered dietitian.

Treatment group received the low- calorie diet including (30g/day) rice bran oil.

ELIGIBILITY:
Inclusion Criteria:

* hyperlipidemia

Exclusion Criteria:

* pregnancy and lactation
* cardiovascular disease
* diabetes

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
LDL, HDL, Cholesterol,Triglyceride(mg/dl) | 30 days
  enzymatic reagents

SECONDARY OUTCOMES:
BMI (Kg/m2) | Baseline and 4 weeks after intervention
  weight/(height)2
WHR (Ratio) | Baseline and 4 weeks after intervention
  Waist(Cm)/Hip(Cm)

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Noroozi, PhD, Principal Investigator — Qazvin University of Medical Sceience
Locations (1):
- Qazvin University of Medical Sciences, Qazvin, Qazvin Province, Iran